CLINICAL TRIAL: NCT01879488
Title: Effect of Ventilation Mode on Lung Deposition of a Radiolabeled Aerosol During Mechanical Ventilation: Barometric Versus Volumetric
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AeroVent-01
Record Dates: First submitted 2013-06-10; First posted 2013-06-17 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Post-operative Neurosurgery
Keywords: Aerosol; Lung deposition; Mechanical ventilation

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Nebulization during pressure support ventilation (Active Comparator): Patients ventilated in pressure support mode during nebulization
  Interventions: Drug: technetium-99m - Diethylenetriaminepentaacetic acid; Device: Vibrating-mesh nebulizer; Other: Gamma scintigraphy; Other: Preoperative spirometry
- Nebulization during volume assist control mode (Active Comparator): Patients ventilated in volume assist control mode during nebulization
  Interventions: Drug: technetium-99m - Diethylenetriaminepentaacetic acid; Device: Vibrating-mesh nebulizer; Other: Gamma scintigraphy; Other: Preoperative spirometry

INTERVENTIONS:
Drug: technetium-99m - Diethylenetriaminepentaacetic acid
Device: Vibrating-mesh nebulizer
Other: Gamma scintigraphy
Other: Preoperative spirometry

SUMMARY:
Controlling the respiratory pattern of mechanically ventilated patients in volume control mode is recommended during nebulization. No studies looked into conditions of nebulization during assisted mechanical ventilation to define the optimal nebulization technique and its effect on pulmonary deposition.

The aim of this study is to analyse the effect of ventilation mode (barometric versus volumetric) on deposition by planar scintigraphy during mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Invasive mechanical ventilation
* Healthy lungs

Exclusion Criteria:

* Change of ventilation mode during nebulization

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2013-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Pulmonary deposition | Immediately after nebulization by imaging assessment, an expected average of 30 minutes

SECONDARY OUTCOMES:
Penetration index | Immediately after nebulization by imaging assessment, an expected average of 30 minutes
Mechanical ventilation settings | During nebulisation time, an expected average of 15 minutes
Lung function | Preoperative assessment, the day before inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-François Laterre, Study Chair — Head of Intensive Care Unit, Cliniques Universitaires Saint-Luc
Locations (1):
- Cliniques Universitaires Saint-Luc, Brussels, Belgium

REFERENCES:
- [Derived] Dugernier J, Reychler G, Wittebole X, Roeseler J, Depoortere V, Sottiaux T, Michotte JB, Vanbever R, Dugernier T, Goffette P, Docquier MA, Raftopoulos C, Hantson P, Jamar F, Laterre PF. Aerosol delivery with two ventilation modes during mechanical ventilation: a randomized study. Ann Intensive Care. 2016 Dec;6(1):73. doi: 10.1186/s13613-016-0169-x. Epub 2016 Jul 22. PMID 27447788